CLINICAL TRIAL: NCT04388657
Title: Study of the Prevalence of Deep Vein Thrombosis in Patients Hospitalized in Intensive Care for Acute Respiratory Failure Linked to Pneumonia Documented With SARS-COV2
Brief Title: COVID-19, bLOod Coagulation and Thrombosis
Acronym: CLOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Hôpital Privé Jacques Cartier, service réanimation Dr Bougouin (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A00
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: COVID; Embolism and Thrombosis; Pneumonia, Viral
MeSH Terms: conditions — Embolism and Thrombosis; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid Intensive arm: Patients included in intensive care admission by one of the principal investigators from the 3 selectioned centers.
  Interventions: Diagnostic Test: Echo-Doppler

INTERVENTIONS:
Diagnostic Test: Echo-Doppler — Utrasound Doppler of the lower limbs

SUMMARY:
Coronavirus 2 (SARS-CoV2) has been identified as the pathogen responsible for severe acute respiratory syndrome associated with severe inflammatory syndrome and pneumonia (COVID-19).

Haemostasis abnormalities have been shown to be associated with a poor prognosis in these patients with this pneumonia. In a Chinese series of 183 patients, the hemostasis balance including thrombin time, fibrinogenemia, fibrin degradation products and antithrombin III were within normal limits. Only the D-Dimer assay was positive in the whole cohort with an average rate of 0.66 µg / mL (normal <50 µg / mL). These hemostasis parameters were abnormal mainly in patients who died during their management; the levels of D-dimers and fibrin degradation products were significantly higher while the antithrombin III was reduced. The findings on the particular elevation of D-dimers in deceased patients as well as the significant increase in thrombin time were also reported in another series. Higher numbers of pulmonary embolisms have been reported in patients with severe form of SARS-COV2 (data in press).

This research is based on the hypothesis that the existence of deep vein thrombosis (DVT) could make it possible to screen patients at risk of pulmonary embolism and to set up a curative anticoagulation.

The main objective is to describe the prevalence of deep vein thrombosis in patients hospitalized in intensive care for acute respiratory failure linked to documented SARS-COV2 pneumonia, within 24 hours of their admission.

DETAILED DESCRIPTION:
Coronavirus 2 (SARS-CoV2) has been identified as the pathogen responsible for severe acute respiratory syndrome associated with severe inflammatory syndrome and pneumonia (COVID-19).

Described at the end of 2019 in China, the pandemic sees the number of patients increasing worldwide, Europe being still in the ascending phase of the epidemic and the American continent at the very beginning of it.

Haemostasis abnormalities have been shown to be associated with a poor prognosis in these patients with this pneumonia. In a Chinese series of 183 patients, the hemostasis balance including thrombin time, fibrinogenemia, fibrin degradation products and antithrombin III were within normal limits. Only the D-Dimer assay was positive in the whole cohort with an average rate of 0.66 µg / mL (normal <50 µg / mL). These hemostasis parameters were abnormal mainly in patients who died during their management; the levels of D-dimers and fibrin degradation products were significantly higher while the antithrombin III was reduced. The findings on the particular elevation of D-dimers in deceased patients as well as the significant increase in thrombin time were also reported in another series. Higher numbers of pulmonary embolisms have been reported in patients with severe form of SARS-COV2 (data in press).

This research is based on the hypothesis that the existence of deep vein thrombosis (DVT) could make it possible to screen patients at risk of pulmonary embolism and to set up a curative anticoagulation. This is all the more important since the occurrence of a pulmonary embolism can clearly worsen the right ventricular failure possibly observed during mechanical ventilation in these patients.

Cohort study, non-interventional, multicentric, prospective, non-comparative, longitudinal.

The main objective of the research is to describe the prevalence of deep vein thrombosis in patients hospitalized in intensive care for acute respiratory failure linked to documented SARS-COV2 pneumonia, within 24 hours of their admission.

The secondary objectives of the research are:

* Identify the factors associated with the existence of deep vein thrombosis
* Describe the relationship between the inflammatory status of patients on admission and the existence of DVT during follow-up.
* Describe the relationship between the results of the hemostasis assessment and the existence of deep vein thrombosis during follow-up.
* Describe the relationship between a right ventricular failure or dysfunction during follow-up and the existence of DVT.
* Describe the relationship between mortality and the existence of DVT, within 28 days of the patient's admission to intensive care or intensive care. Describe the lung parenchyma if a CT scan is performed

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age with no upper age limit.
* Patient admitted to intensive care or intensive care for pneumonia linked to SARS-COV2 (diagnosed on positive PCR or chest CT and anamnesis)
* Affiliated patient or beneficiary of a social security scheme
* Patient having been informed and not objecting to the use of their data in the context of this research.

Exclusion Criteria:

* Pregnant, lactating or parturient woman
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient admitted in intensive care
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with one or more DVTs. | 28 days
  The primary outcome measure will be the percentage of patients with one or more DVTs from a lower extremity ultrasound scan.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Ambroise Paré, Boulogne-Billancourt, IDF
  - Hôpital Privé Jacques Cartier, Massy, IDF
  - Centre Cardiologique du Nord, Saint-Denis, IDF

IPD SHARING:
Plan to Share IPD: Undecided